CLINICAL TRIAL: NCT04123977
Title: Evaluation of Patient Analgesia After Bloc Serratus for the Management of Thoracic Trauma
Brief Title: Evaluation of Patient Analgesia After Bloc Serratus
Acronym: TraumaThorax
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7406
Record Dates: First submitted 2019-10-03; First posted 2019-10-11 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Thorax Traumas
Keywords: thorax trauma; head injury; Multi-modal analgesia; Paravertebral block; Thoracic epidural; Serratus Block
MeSH Terms: conditions — Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Thorax traumas are very common in severe traumatology, including road accidents, representing the second most frequent site (after head injury, according to the FIRST study). These thoracic lesions are the cause of many complications (pneumothorax, hemothorax, lung infections, atelectasis).

The national recommendations recommend the use of multi-modal analgesia with the use of regional loco anaesthesia for pain management and prevention of respiratory complications, including infectious complications. The loco-regional anaesthesia of choice is thoracic epidural or paravertebral block, but these techniques are not without risks, and are contraindicated in many situations (severe head trauma, patient under curative anticoagulation, pelvic trauma...).

The anterior Serratus block appears to be a quality localoregional anaesthesia in thoracic surgery, and a few cases in the literature have shown an interest in severe traumatology.

The investigators perform this anterior Serratus block almost systematically in patients with thoracic trauma in the Hautepierre surgical intensive care unit.

ELIGIBILITY:
Inclusion criteria:

* Adult patient (≥18 years old)
* Gender (Male and Female)
* Patient hospitalised in surgical intensive care or continuous trauma care with thorax trauma who received anterior Serratus block analgesia from January 1, 2018 to February 28, 2019
* Patient who has given his consent to the reuse of his data for the purposes of this research

Criteria for non-inclusion:

* Patient who has expressed opposition to participating in the study
* Impossibility of giving the subject informed information (difficulties in understanding the subject,...)
* Subject under the protection of justice
* Subject under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient hospitalised in surgical intensive care or continuous trauma care with thorax trauma who received anterior Serratus block analgesia from January 1, 2018 to February 28, 2019
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Retrospective analysis of analgesia after Bloc serratus | Files analysed retrospectily from January 1st, 2018 to February 28, 2019 will be examined

CONTACTS AND LOCATIONS:
Overall Officials: Julien POTTECHER, MD, PhD, Study Director — University Hospital, Strasbourg, France
Locations (1):
- Service de Réanimation chirurgicale_ Hôpital de Hautepierre, Strasbourg, France